CLINICAL TRIAL: NCT01031615
Title: Evaluation of the Child and Family Traumatic Stress Intervention
Acronym: CFTSI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Carla S. Stover/Assistant Professor, Yale University School of Medicine Child Study Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0504027679; SAMHSA U79SM54318 (Other Grant/Funding Number: SAMHSA U79SM54318)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: School age children and adolescents exposed to a potentially traumatic event
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Child and Family Traumatic Stress Interv (Experimental): 4-session secondary prevention model that focuses on family communication about symptoms of a child aged 7-16.
  Interventions: Behavioral: Child and Family Traumatic Stress Interv (CFTSI)
- Psychoeducational Comparison (Active Comparator): 4-sessions focused on individual child using psychoeducation and relaxation skills
  Interventions: Behavioral: Psychoeducational Comparison

INTERVENTIONS:
Behavioral: Child and Family Traumatic Stress Interv (CFTSI) — 4 sessions involving both the target child and a parent/caregiver
  Arms: Child and Family Traumatic Stress Interv
Behavioral: Psychoeducational Comparison — 4 individually focused sessions including psychoeducation and relaxation.
  Arms: Psychoeducational Comparison

SUMMARY:
The purpose of this study is to determine the efficacy of the Child and Family Traumatic Stress Intervention (CFTSI) in preventing the development of Posttraumatic Stress Disorder (PTSD) when implemented within 30 days of a potentially traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Youth exposed to a potentially traumatic event within the last 30 days who have one new symptom on the Posttraumatic Checklist (PCL)

Exclusion Criteria:

* Already receiving mental health treatment
* Autism or Developmental Disability
* Diagnosed with psychosis or bipolar disorder
* Non-english speaking

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2005-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
UCLA Posttraumatic Reaction Index (PTSD-RI) | 3 months post-intervention

SECONDARY OUTCOMES:
Trauma Symptom Checklist for Children (TSCC) | 3 Months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Steven Berkowitz, M.D., Study Director — University of Pennsylvania
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Berkowitz SJ, Stover CS, Marans SR. The Child and Family Traumatic Stress Intervention: secondary prevention for youth at risk of developing PTSD. J Child Psychol Psychiatry. 2011 Jun;52(6):676-85. doi: 10.1111/j.1469-7610.2010.02321.x. Epub 2010 Sep 24. PMID 20868370